CLINICAL TRIAL: NCT04420078
Title: Brugada Ablation of VF Substrate Ongoing MultiCenter Registry
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Pacific Rim Electrophysiology Research Institute (Other)
Collaborators: University Hospital, Bordeaux (Other); University of Tsukuba (Other); University of London (Other); University of Amsterdam (Other); Ogaki Municipal Hospital (Unknown); Indiana University (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: BRAVO Registry
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CA BrS: Symptomatic BrS patients who underwent catheter ablation of the BrS/VF substrate
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — Ventricular fibrillation substrate

SUMMARY:
Current treatment of high-risk Brugada Syndrome (BrS) patients (pts) with recurrent VF is limited. Catheter ablation (CA) has been performed for BrS but a large study with long-term outcomes of CA in BrS ablation are lacking.

DETAILED DESCRIPTION:
Brugada syndrome (BrS) patients who undergo BRS substrate ablations from tertiary centers for catheter ablations of complex arrhythmias from three continents - Asia, Europe and North America - are registered in a common database. The investigators exclude patients who were lost to follow up in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Brugada Syndrome patients who had undergone catheter ablation of the arrhythmogenic substrates.

Exclusion Criteria:

* Patients who will not commit to regular follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have positive Brugada ECG pattern and have underwent catheter ablation of VF substrates prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Death | 3 years
  Expiration, unrelated to procedure
ICD Therapy for VT/VF | 3 years
  Electrical therapy delivered through device for termination of VF episodes

SECONDARY OUTCOMES:
Inappropriate ICD Therapy | 3 years
  Caused by lead sensing or programming errors
Normalization of Brugada ECG pattern | 3 years
  ECG pattern is normal sinus rhythm after catheter ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Rim Electrophysiology Research Institute, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
All data published will be deindentified

REFERENCES:
- [Derived] Nademanee K, Chung FP, Sacher F, Nogami A, Nakagawa H, Jiang C, Hocini M, Behr E, Veerakul G, Jan Smit J, Wilde AAM, Chen SA, Yamashiro K, Sakamoto Y, Morishima I, Das MK, Khongphatthanayothin A, Vardhanabhuti S, Haissaguerre M. Long-Term Outcomes of Brugada Substrate Ablation: A Report from BRAVO (Brugada Ablation of VF Substrate Ongoing Multicenter Registry). Circulation. 2023 May 23;147(21):1568-1578. doi: 10.1161/CIRCULATIONAHA.122.063367. Epub 2023 Mar 24. PMID 36960730